CLINICAL TRIAL: NCT04966065
Title: Evaluation of the Parietex TM Parastomal No Hole Mesh for Repair of Parastomal Hernias in End-colostomieswith a Laparoscopic Modified Sugarbaker Technique in a Prospective Multicenter International Observational Study
Brief Title: Evaluation of the Parietex TM Parastomal No Hole Mesh for Repair of Parastomal Hernias in End-colostomies
Acronym: PHARAO
Status: Terminated | Type: Observational
Why Stopped: too slow patiënts recruitment
Sponsor: University Hospital, Ghent (Other)
Collaborators: Algemeen Ziekenhuis Maria Middelares (Other); University of Wuerzburg (Other); Universitaire Ziekenhuizen KU Leuven (Other); Bispebjerg Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2015_0164
Record Dates: First submitted 2021-07-07; First posted 2021-07-19 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Parastomal Hernia
Keywords: ostomy; hernia; parastomal; sugarbaker
MeSH Terms: conditions — Hernia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Parietex Parastomal mesh — Laparoscopic Modified Sugarbaker technique for repair of parastomal hernias in end-colostomies

SUMMARY:
Short Title: PHARAOH study: LAPAROSCOPIC PARASTOMAL HERNIA REPAIR WITH A NO HOLE MESH.

Objectives:

Evaluation of operative complications, colostomy function, Quality of Life and recurrence rate after laparoscopic repair of parastomal hernias in end-colostomies with a ParietexTM Parastomal No Hole mesh.

Principle Investigators:

Prof. Dr. Frederik Berrevoet, University Hospital Ghent Dr. Filip Muysoms, AZ Maria Middelares Ghent

Patient selection:

Adult consecutive patients, men or women, aged above 18, planned for primary elective laparoscopic hernia repair of an end-colostomy. A logbook will be kept of adult patients undergoing a parastomal hernia repair in the participating centers during the study period that are not entered in the study, including the reason for non inclusion. A total of 100 patients will be included during 24 months or until the sample size has been reached.

Exclusion criteria: previous repair of a parastomal hernia at the same site, emergency operations, open parastomal hernia repair, parastomal hernias at an ileostomy or an ileal conduit stoma, loop colostomies, patients under the age of 18 years, pregnant women, ASA score 4 or more, no informed consent of the patient, patients unable to complete the stoma Quality of Life assessment.

Primary Endpoint:

Evolution of Quality of Life with the Stoma-QoL score assessment of patients: preoperatively, at 1 month, 12 months and 24 months postoperatively.

Secondary Endpoints:

Quality of Life of the patients with the EuraHS QoL score: preoperatively, at 1 month, 12 months and 24 month postoperatively. Recurrence rate at 12 and at 24 months postoperatively evaluated by clinical examination and if available computer tomography. Intra-operative and post-operative complications, post-operative hospital stay, operation time.

DETAILED DESCRIPTION:
Primary Endpoint:

Evolution of Quality of Life with the Stoma-QoL score assessment of patients: preoperatively, at 1 month, 12 months and 24 months postoperatively.

Secondary Endpoints:

Quality of Life of the patients with the EuraHS QoL score: preoperatively, at 1 month, 12 months and 24 month postoperatively. Recurrence rate at 12 and at 24 months postoperatively evaluated by clinical examination and if available computer tomography. Intra-operative and post-operative complications, post-operative hospital stay, operation time.

ELIGIBILITY:
Inclusion Criteria:

- adult patients, planned for primary elective laparoscopic hernia repair of an end-colostomy.

Exclusion Criteria:

* previous repair of a parastomal hernia at the same site
* emergency operations
* open parastomal hernia repair
* parastomal hernias at an ileostomy or an ileal conduit stoma
* loop colostomies
* patients under the age of 18 years
* pregnant women
* ASA score 4 or more
* no informed consent of the patient
* patients unable to complete the stoma Quality of Life assessment

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 100 adult patients, men or women, aged above 18, planned for primary elective laparoscopic hernia repair of an end-colostomy.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2016-03-14 (Actual); Primary Completion 2018-09-24 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of the QoL with the Stomy-QoL score assessment | 24 months
  Evaluation of the QoL with the Stomy-QoL score assessment of patients preop, at 1 month, 12 months and 24 months postoperatively

SECONDARY OUTCOMES:
Recurrence rate | 24 months
  Evaluation of the recurrence rates after surgical repair
Peri-operative complications | 6 months
  All intra- and postoperative complications involving the surgical procedure

CONTACTS AND LOCATIONS:
Overall Officials: Frederik Berrevoet, MD, PhD, Principal Investigator — University Ghent
Locations (1):
- Ghent University Hospital, Ghent, East Flanders, Belgium

IPD SHARING:
Plan to Share IPD: No